CLINICAL TRIAL: NCT02051621
Title: Isolated Atrial Fibrillation Ablation in Patients With Isolated Atrial Flutter
Brief Title: Therapy of Atrial Flutter by Afib Ablation
Acronym: TripleA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rostock (Other)
Collaborators: Biosense Webster, Inc. (Industry); Medtronic (Industry)
Responsible Party: Principal Investigator, Dietmar Baensch, Professor Dr. med., University of Rostock
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A201070
Record Dates: First submitted 2013-12-03; First posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: pulmonary vein isolation; isthmus ablation; recurrence
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Recurrence | interventions — Anti-Arrhythmia Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cavo-tricuspid-isthmus-ablation (Active Comparator): Ablation of atrial flutter
  Interventions: Procedure: Cavo-tricuspid-isthmus-ablation
- Pulmonary vein isolation (Active Comparator): pulmonary vein isolation
  Interventions: Procedure: Pulmonary vein isolation
- Antiarrhythmic drug (Active Comparator): Medical treatment of atrial flutter with either class I antiarrhythmics (flecainide (Tambocor ®) 100 mg twice daily or propafenone (Rytmonorm ®) up to 150 mg 3 times daily) or amiodarone (Cordarex®) 200 mg daily
  cardioversion as needed
  Interventions: Drug: Antiarrhythmic drug

INTERVENTIONS:
Drug: Antiarrhythmic drug — medical treatment of atrial flutter with either flecainide (Tambocor ®) 100 mg twice daily, propafenone (Rytmonorm ®) up to 150 mg 3 times daily) or amiodarone (Cordarex®) 200 mg daily electrical cardioversion as needed
  Other Names: medical treatment of atrial flutter
  Arms: Antiarrhythmic drug
Procedure: Cavo-tricuspid-isthmus-ablation — irrigated radiofrequency (RF)-ablation of the cavo-tricuspid-isthmus catheter used: Thermocool R (F-type), Biosense Webster, Diamond Bar, CA, USA
  Other Names: Ablation of atrial flutter
  Arms: Cavo-tricuspid-isthmus-ablation
Procedure: Pulmonary vein isolation — pulmonary vein angiography followed by antral pulmonary vein isolation using 3D-electroanatomical Mapping mapping system: Carto 3 (Biosense Webster, Diamond Bar, CA, USA) catheter used for irrigated RF-ablation: Navistar Thermocool R (D, E or F-type according to atrial dimensions), Biosense Webster, Diamond Bar, CA, USA
  Arms: Pulmonary vein isolation

SUMMARY:
Ablation of the cavotricuspid isthmus (CTI) in the right atrium is currently the therapy of choice for the treatment of typical atrial flutter (3,4). It is a curative approach and has a high success rate (5). It has been recognized that patients with typical atrial flutter often complain of atrial fibrillation (1,2). Current clinical and experimental studies confirm the close relationship between atrial flutter (AFL) and atrial fibrillation (AF) and raise a question, if both arrhythmias are different forms of a common electrical phenomenon with atrial fibrillation being the underlying clinical problem (6).

DETAILED DESCRIPTION:
Current clinical and experimental studies confirm the close relationship between atrial flutter (AFlut) and atrial fibrillation (Afib). After initiation of Afib this may organize under special intrinsic conditions or due to antiarrhythmic medication to AFlut so Afib may be supposed the underlying arrhythmia. Therefore after successful ablation of AFlut this reentrant circuit is not longer possible and Afib persists. After new occurrence of Afib a long diagnostic and therapeutic marathon begins with AF ablation at the end of all therapeutic efforts. This double burden for the patient and the health system can probably be avoided by directly and effectively treating the underlying arrhythmia AF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with- in 12-Channel-ECG documented atrial tachycardia suggestive of typical isthmus dependent atrial flutter
* > 21 years

Exclusion Criteria:

* - AFL as secondary to an accessory pathway
* Antiarrhythmic treatment for AF
* AF
* Previous AF ablation
* Dilatation of left atrium > 6 cm
* Cardiac surgery less < 3 weeks
* Congenital heart disease
* Cardiac ischemia or coronary artery disease that needs intervention
* Life expectancy less than 2 years

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-08; Primary Completion 2015-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Number or patients with a recurrence of any atrial arrhythmia | 2 years
  Number (percentage) of patients with any atrial arrhythmia lasting longer than 30 s after ablation assessed by implantable loop recorder or 7-day-holter-ECG: AFL after AF ablation compared to the AFL ablation group and AF in both ablation groups

SECONDARY OUTCOMES:
Number of patients with atrial flutter recurrence | 2 years
  Number (percentage) of patients with any AFL episode after ablation or under medical therapy assessed by implantable loop recorder or 7-day-holter-ECG, compared between all 3 interventions (medical treatment vs. AFL Ablation vs. AF ablation)

CONTACTS AND LOCATIONS:
Overall Officials: Dietmar Baensch, PhD, MD, Principal Investigator — University Medical Centre Rostock
Locations (1):
- Universitiy Medical Centre Rostock, Rostock, Germany

REFERENCES:
- [Derived] Schneider R, Lauschke J, Tischer T, Schneider C, Voss W, Moehlenkamp F, Glass A, Diedrich D, Bansch D. Pulmonary vein triggers play an important role in the initiation of atrial flutter: Initial results from the prospective randomized Atrial Fibrillation Ablation in Atrial Flutter (Triple A) trial. Heart Rhythm. 2015 May;12(5):865-71. doi: 10.1016/j.hrthm.2015.01.040. Epub 2015 Jan 28. PMID 25638698